CLINICAL TRIAL: NCT01874327
Title: Joint Engagement in Infants at Risk for ASD: Integrating Treatment With Biomarkers
Brief Title: Biomarkers of Developmental Trajectories and Treatment in Autism Spectrum Disorder (ASD)
Acronym: BabyJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-000607
Record Dates: First submitted 2012-10-28; First posted 2013-06-11 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Children at Risk for ASD

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baby JASPER (Active Comparator): This classroom will spend the majority of the time focusing on social-communication goals
  Interventions: Behavioral: Baby JASPER
- Standard Baby Classroom (Active Comparator): This classroom will focus more heavily on developing motor and cognitive skills
  Interventions: Behavioral: Standard Baby Classroom

INTERVENTIONS:
Behavioral: Baby JASPER — Intervention focuses on core deficits of joint attention, play, engagement, and regulation embedded within AEPS curriculum
  Arms: Baby JASPER
Behavioral: Standard Baby Classroom — Assessment, Education and Programming System (AEPS) for Infants and Children curriculum focused on early developmental milestones in fine and gross motor, cognitive, adaptive and social areas
  Arms: Standard Baby Classroom

SUMMARY:
The study will evaluate the efficacy of a novel intervention implemented in a classroom setting aimed at improving joint attention and joint engagement skills with infants who are at risk of developing an Autism Spectrum Disorder.

DETAILED DESCRIPTION:
The proposed intervention adapts a parent-mediated intervention that successfully improved outcomes in toddlers with autism. The intervention model (a) targets the foundations of social-communication (joint attention, imitation, play), (b) uses naturalistic strategies to increase the rate and complexity of social-communication and (c) includes parents as implementers of the intervention to promote generalization across settings and activities and to ensure maintenance over time.

In addition to testing the primary effects of this early intervention on the developmental outcomes of children with signs of autism, we will examine whether this method is superior to an early intervention focused on global infant development. Because brain development occurs rapidly in infants and toddlers, we will use high density EEG to investigate (1) biomarkers of change in these infants as a result of intervention and (2) biomarkers predicting response to treatment, with focus on the neural correlates of social attention and learning from joint engagement.

Study Aims:

AIM 1: To examine the effects of the experimental intervention (Baby JASPER) on primary (joint attention) and secondary outcomes (receptive language, play, symbol-infused joint engagement and parent use of social communication support strategies).

AIM 2: To examine maintenance and generalization of the effects of the experimental intervention on children and their parents.

AIM 3: To examine electrophysiological biomarkers of change with treatment as well as predictors of social communication outcomes in children after intervention.

AIM 4 (exploratory): To examine the effect of potential child level and parent level moderators on the primary and secondary outcomes of the study across the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Have elevated scores on the ADOS-Toddler version and clinical concern from professional (Pediatrician, Psychologist, etc). Because of the young age of children, we expect to intervene with children who do not yet have a diagnosis of ASD but may only show some risk by virtue of elevated scores on the ADOS-T.
* Have a parent available for parent-mediated sessions 2 times per week in the classroom
* Do not have seizures
* Do not have associated sensory or physical disorders
* Are not co-morbid with other syndromes or diseases

Exclusion Criteria:

* Other co-morbid syndromes or diseases
* Seizure activity
* Other sensory or physical disorders

Ages: 12 Months to 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Assessing change in Parent Child Interaction (PCX) throughout the diverse time points. | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)
  10 minute unstructured free play assessment with caregiver and child measuring change over the duration of the study.

SECONDARY OUTCOMES:
Autism Diagnostic Observation Schedule Toddler module (ADOS-T) | Prior to treatment commencing (Study Entry) and 10 months post treatment exit
  Semi-structured, standardized assessment of communication, social interaction, play and imaginative use of materials
Imitation Task | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)
Vineland Adaptive Behavior Scales (VABS) | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)
EEG/Event Related Potential (ERP) | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)
Mullen Scales of Early Learning (MSEL) | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)
Early Social Communication Scales (ESCS) | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)
Structured Play Assessment (SPA) | Prior to treatment commencing (Study Entry), within treatment (3 and 6 weeks post entry), Exit (8-10 weeks post entry), and three further follow ups (2 months post exit, 4 months post exit and 10 months post exit)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institue, Los Angeles, California, United States

REFERENCES:
- [Background] Abidin, R. R. (1983). Parenting Stress Index manual. Charlottesville, VA: Pediatric Psychology Press.
- [Background] Adamson LB, Bakeman R, Deckner DF. The development of symbol-infused joint engagement. Child Dev. 2004 Jul-Aug;75(4):1171-87. doi: 10.1111/j.1467-8624.2004.00732.x. PMID 15260871
- [Background] Akhtar N, Dunham F, Dunham PJ. Directive interactions and early vocabulary development: the role of joint attentional focus. J Child Lang. 1991 Feb;18(1):41-9. doi: 10.1017/s0305000900013283. PMID 2010504
- [Background] Arnold, S. D., Elliot, M., Storoschuk, S., Pickles, A., Hellriegel, C., & Lord, C. (1993) Social directedness and prelinguistic vocalization in autism. Paper presented at the meeting of the American Academy of Child and Adolescent Psychiatry, San Antonio, TX.
- [Background] Bakeman R, Adamson LB. Coordinating attention to people and objects in mother-infant and peer-infant interaction. Child Dev. 1984 Aug;55(4):1278-89. PMID 6488956
- [Background] Barnes S, Gutfreund M, Satterly D, Wells G. Characteristics of adult speech which predict children's language development. J Child Lang. 1983 Feb;10(1):65-84. doi: 10.1017/s0305000900005146. No abstract available. PMID 6841502
- [Background] Baron-Cohen S. The autistic child's theory of mind: a case of specific developmental delay. J Child Psychol Psychiatry. 1989 Mar;30(2):285-97. doi: 10.1111/j.1469-7610.1989.tb00241.x. PMID 2523408
- [Background] Baron-Cohen, S. (1993). From attention-goal psychology to belief-desire psychology: The development of a theory of mind and its dysfunction. In S. Baron-Cohen, H. Tager-Flusberg, & D. J. Cohen (Eds.), Understanding other minds: Perspectives from autism, Oxford, UK: Oxford University Press.
- [Background] Brereton, A., & Tonge, B. (2005). Pre-schoolers with autism: An education and skills training programme for parents. London, UK: Jessica Kingsley Publishers.
- [Background] Brown, R. (1973). A first language: The early stages. Cambridge, MA: Harvard University Press.
- [Background] Bruner, J.S. (1974/75). From communication to language: A psychological perspective. Cognition, 3, 255-287.
- [Background] Bryk, A., & Raudenbush, S. (1992). Hierarchical linear models: Applications and data analysis methods. Newborn Park, CA: Sage.
- [Background] Cross, T. G. (1977). Mother's speech adjustments: The contribution of selected child listener variables. In C. E. Snow and C. A. Ferguson (Eds.), Talking to children: Language input and acquisition. Cambridge: Cambridge University Press.
- [Background] Curcio F. Sensorimotor functioning and communication in mute autistic children. J Autism Child Schizophr. 1978 Sep;8(3):281-92. doi: 10.1007/BF01539631. PMID 690064
- [Background] D'Amico EJ, Neilands TB, Zambarano R. Power analysis for multivariate and repeated measures designs: a flexible approach using the SPSS MANOVA procedure. Behav Res Methods Instrum Comput. 2001 Nov;33(4):479-84. doi: 10.3758/bf03195405. PMID 11816450
- [Background] Dawson, G., & Galpert, L. (1990). Mother's use of imitative play for facilitating social responsiveness and toy play in young autistic children. Development and Psychopathology, 2, 151-162.
- [Background] Dawson, G., & Osterling, J. (1997). Early intervention in autism: Effectiveness and common elements of current approaches. In Guralnick, M. J. (Ed.), The Effectiveness of Early Intervention: Second Generation Research (pp. 307-326). Balitmore, MD: Brookes.
- [Background] Donnellan, A & Kilman, B. (1986). Behavioral approaches to social skill development in autism: Strengths, misapplications, and alternatives. In E. Schopler & G. Mesibov (Eds.), Social behavior in autism, (pp. 213-236). New York: Plenum Press.
- [Background] Harding, C. G. (1983). Setting the stage for language acquisition: Communication in the first year. In R. M. Golinkoff (Ed.), The transition from prelinguistic to linguistic communication. Hillsdale, NJ: Erlbaum.
- [Background] Harris S, Kasari C, Sigman MD. Joint attention and language gains in children with Down syndrome. Am J Ment Retard. 1996 May;100(6):608-19. PMID 8735574
- [Background] Hobson, R. P. (1989). On sharing experiences. Development and Psychopathology, 1, 197-203.
- [Background] Lovaas OI. Behavioral treatment and normal educational and intellectual functioning in young autistic children. J Consult Clin Psychol. 1987 Feb;55(1):3-9. doi: 10.1037//0022-006x.55.1.3. No abstract available. PMID 3571656
- [Background] Kaiser, A., Yoder, P., & Keetz, A. (1992). Evaluating milieu teaching. In S. Warren & J. Reichle (Eds.), Causes and effects in communication and language intervention. (pp. 9-47). Baltimore, MD: Brookes.
- [Background] Kanner L. Autistic disturbances of affective contact. Acta Paedopsychiatr. 1968;35(4):100-36. No abstract available. PMID 4880460
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Kasari C, Mundy P, Yirmiya N, Sigman M. Affect and attention in children with Down syndrome. Am J Ment Retard. 1990 Jul;95(1):55-67. PMID 2143659
- [Background] Kasari C, Sigman M. Linking parental perceptions to interactions in young children with autism. J Autism Dev Disord. 1997 Feb;27(1):39-57. doi: 10.1023/a:1025869105208. PMID 9018581
- [Background] Kasari C, Sigman MD, Baumgartner P, Stipek DJ. Pride and mastery in children with autism. J Child Psychol Psychiatry. 1993 Mar;34(3):353-62. doi: 10.1111/j.1469-7610.1993.tb00997.x. PMID 8463373
- [Background] Kasari C, Sigman M, Mundy P, Yirmiya N. Caregiver interactions with autistic children. J Abnorm Child Psychol. 1988 Feb;16(1):45-56. doi: 10.1007/BF00910499. PMID 2966189
- [Background] Kasari C, Sigman M, Mundy P, Yirmiya N. Affective sharing in the context of joint attention interactions of normal, autistic, and mentally retarded children. J Autism Dev Disord. 1990 Mar;20(1):87-100. doi: 10.1007/BF02206859. PMID 2139025
- [Background] Kasari, C., Sigman, M., Yirmiya, N., & Mundy, P. (1993). Affective development and communication in children with autism. In A.P. Kaiser & D.B. Gray (Eds.), Enhancing children's communication: Research foundations for intervention (pp. 201-222). New York: Brookes.
- [Background] Kasari, C., Sigman, M., & Yirmiya, N. (1994). Focused and social attention in caregiver-child interactions: A comparison of autistic, mentally retarded and nonretarded children. Development and Psychopathology, 5, 403-414.
- [Background] Kellam SG, Rebok GW, Ialongo N, Mayer LS. The course and malleability of aggressive behavior from early first grade into middle school: results of a developmental epidemiologically-based preventive trial. J Child Psychol Psychiatry. 1994 Feb;35(2):259-81. doi: 10.1111/j.1469-7610.1994.tb01161.x. PMID 8188798
- [Background] Kirk, R.E. (1982). Experimental design: Procedures for the behavioral sciences. (2nd ed). Pacific Grove CA: Brooks/Cole.
- [Background] Koegel RL, Firestone PB, Kramme KW, Dunlap G. Increasing spontaneous play by suppressing self-stimulation in autistic children. J Appl Behav Anal. 1974 Winter;7(4):521-8. doi: 10.1901/jaba.1974.7-521. PMID 4443320
- [Background] Koegel, R., & Koegel, L. (1995). Teaching children with autism. Baltimore: Paul H. Brookes.
- [Background] Lord, C., Rutter, M.D., DiLavore, P. & Risi, S. (2001). Autism diagnostic observation schedule manual. Los Angeles, CA: Western Psychological Services.
- [Background] Lord, C., Storoschuk, S., Rutter, M. & Pickles, A. (1993). Using the ADI-R to diagnose autism in preschool children with autism. Infant Mental Health Journal, 14, 234-252.
- [Background] Loveland KA, Landry SH. Joint attention and language in autism and developmental language delay. J Autism Dev Disord. 1986 Sep;16(3):335-49. doi: 10.1007/BF01531663. PMID 3558291
- [Background] Fenson, L., Dale, P. S., Reznick, J. S., Thal, D., Bates, E., Hartung, J. P., Pethick, S., & Reilly, J. S. (1993). The Macarthur communicative development inventories: User's guide and technical manual. San Diego, CA: Singular Publishing Group.
- [Background] McEachin JJ, Smith T, Lovaas OI. Long-term outcome for children with autism who received early intensive behavioral treatment. Am J Ment Retard. 1993 Jan;97(4):359-72; discussion 373-91. PMID 8427693
- [Background] Miller JF, Chapman RS. The relation between age and mean length of utterance in morphemes. J Speech Hear Res. 1981 Jun;24(2):154-61. doi: 10.1044/jshr.2402.154. PMID 7265928
- [Background] Morales, M., Mundy, P., & Rojas, J. (1998). Following the direction of gaze and language development in 6-month-olds. Infant Behavior & Development, 21, 373-377.
- [Background] Mullen, E. (1989). Infant Mullen Scales of Early Learning. Cranston, RI: T.O.T.A.L. Child, Inc. Mundy, P., & Gomes, A. (1998). Individual differences in joint attention skill development in the second year. Infant Behavior & Development, 21, 469-482.
- [Background] Mundy, P., Kasari, C. & Sigman, M. (1992). Nonverbal communication, affective sharing, and intersubjectivity. Infant Behavior and Development, 15, 377-381.
- [Background] Mundy P, Sigman M, Kasari C. A longitudinal study of joint attention and language development in autistic children. J Autism Dev Disord. 1990 Mar;20(1):115-28. doi: 10.1007/BF02206861. PMID 2324051
- [Background] Mundy, P., Sigman, M. & Kasari, C. (1993). The theory of mind and joint-attention deficits in autism. In S. Baron-Cohen, H. Tager-Flusberg, & D. Cohen (Eds.), Understanding other minds: Perspectives from autism (pp. 181-203). New York: Oxford University Press.
- [Background] Mundy, P., Sigman, M., & Kasari, C. (1994). Nonverbal communication, developmental level and symptom presentation in autism. Development and Psychopathology, 6, 389-401.
- [Background] Mundy P, Sigman M, Ungerer J, Sherman T. Defining the social deficits of autism: the contribution of non-verbal communication measures. J Child Psychol Psychiatry. 1986 Sep;27(5):657-69. doi: 10.1111/j.1469-7610.1986.tb00190.x. PMID 3771682
- [Derived] Sterrett K, Magana MT, Gulsrud A, Paparella T, Kasari C. Predictors of Attrition in a Randomized Trial of a Social Communication Intervention for Infant-Toddlers at Risk for Autism. J Autism Dev Disord. 2023 Aug;53(8):3023-3033. doi: 10.1007/s10803-022-05616-w. Epub 2022 Jun 9. PMID 35678946